CLINICAL TRIAL: NCT06543355
Title: The Acupuncture for Pain, Opioid Use Disorder and Mood (AcuPOM) Study: A Pilot Trial
Brief Title: The Acupuncture for Pain, Opioid Use Disorder and Mood
Acronym: AcuPOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2024-15724; 4RM1DA055437-02 (NIH)
Record Dates: First submitted 2024-08-02; First posted 2024-08-09 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain; Opioid Use Disorder; Mood Change; Opioid Misuse; Opioid-Related Disorders
Keywords: Acupuncture
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Acupuncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- BFA + NADA protocol (Experimental): Modified BFA + NADA treatment, twice per week over 4 weeks for a total of 8 treatments at the clinic. All participants will also have the small seeds placed to facilitate at-home acupressure treatment
  Interventions: Device: Modified Battlefield Acupuncture + National Acupuncture Detoxification Association protocol

INTERVENTIONS:
Device: Modified Battlefield Acupuncture + National Acupuncture Detoxification Association protocol — The delivery of modified BFA + NADA will be administered in a setting designed to ensure that patients are comfortable, with their backs well-supported. With regards to needling technique, participants' ears will be cleaned, and sterile acupuncture needles will be placed on the BFA or NADA points, using proper technique. Auricular acupuncture needles are thin, between 0.12 - 0.18mm, and are less than 1 inch long. The needles will remain in the ear until the session is complete. On the alternative ear, seeds are another modality of auricular acupuncture treatment that will be used. Seeds are comprised of small circular balls comprised of a natural plant, no more than 1.5 mm diameter size. The seeds are attached to a small piece of adhesive tape and are placed on one's ear. The seeds remain on the ear and the given point can be massaged and stimulated as indicated.

SUMMARY:
The goal of this study is to determine how patients with chronic pain and opioid use disorder will respond to treatment with acupuncture, including whether there will be any changes in mood (as an exploratory outcome). Results from this study have the potential to inform future studies in patients who would consider using acupuncture as an intervention for their conditions.

DETAILED DESCRIPTION:
In this 4-week pilot study, the feasibility of recruiting a sample of participants in a modified Battlefield Acupuncture + National Acupuncture Detoxification Association (BFA + NADA) protocol will be assessed. Utilizing a novel BFA (Battlefield Acupuncture) plus a NADA (National Acupuncture Detoxification Association) protocol, approximately 20 participants with chronic pain and Opioid Use Disorder (OUD), receiving Methadone through an Opioid Treatment Program (OTP) at Montefiore Medical Center, will be recruited. Each participant will receive a modified BFA + NADA treatment, twice per week over 4 weeks for a total of 8 treatments at the clinic. All participants will also have the small seeds placed to facilitate at-home acupressure treatment. In this feasibility study, the investigator team will collect feasibility data from each participant at every session over the course of 4 weeks. Feasibility outcomes are defined in the Outcome Measures of this registration. As part of the study, the following will also be monitored to explore preliminary efficacy: (1) pain intensity and physical functioning, (2) opioid cravings and substance use, and (3) mood, insomnia, and stress. The research team will conduct surveys assessing pain, physical functions, the changes in stress, mood, insomnia and psychological changes at baseline, and before and after every treatment. These will all be exploratory as this is a feasibility study.

Note: Following discussions with the Principal Investigator and Sponsor this study was re-categorized as a feasibility study.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old,
2. English proficiency;
3. receiving methadone treatment at an OTP through the Montefiore network for at least 12 weeks, with no dose change in 14 days to ensure treatment stability;
4. chronic pain of at least moderate pain severity (score of at least 4 on the Pain, Enjoyment of Life and General Activity (PEG) scale);
5. willingness to participate in all study components; and
6. ability to provide informed consent

Exclusion Criteria:

1. Have pending surgery or invasive pain management procedure;
2. Have a pending or planned relocation;
3. have an acutely or exacerbation of psychotic, suicidal, or homicidal conditions that preclude the ability to participate; and
4. pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Feasibility - Percentage Consented | During the informed consent process, prior to the intervention
  The percentage of total participants screened who have been consented will be calculated and reported.
Feasibility - Percentage Retained | Upon completion of the study, up to four weeks
  The percentage of total participants consented who complete the study will be calculated and reported.
Adherence to acupuncture treatments | At 0, 2, and 4 week study visits, up to four weeks total
  Adherence to acupuncture treatments treatments will also be used to assess feasibility. Adherence the intervention will be defined as the percentage of participants who completed all scheduled acupuncture treatments. Adherence will be successful if participants attend at least 50% of acupuncture treatments.
Acceptability/Satisfaction | Upon completion of the study, up to four weeks
  Acceptability of and Satisfaction with the intervention will be assessed using a single outcome measure, the Patient Global Impression of Change Scale. This scale consists of a single question asking the participant to rate acceptability/satisfaction of the intervention on a seven-point scale ranging from 1 (= very much better) to 7 ( = very much worse). Higher scores are associated with less favorable participant perceptions of the intervention. Group mean scores will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Bayner, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Division of Substance Abuse (DoSA) Wellness Center at Melrose, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dahlhamer J, Lucas J, Zelaya C, Nahin R, Mackey S, DeBar L, Kerns R, Von Korff M, Porter L, Helmick C. Prevalence of Chronic Pain and High-Impact Chronic Pain Among Adults - United States, 2016. MMWR Morb Mortal Wkly Rep. 2018 Sep 14;67(36):1001-1006. doi: 10.15585/mmwr.mm6736a2. PMID 30212442
- [Background] Patel M, Urits I, Kaye AD, Viswanath O. The role of acupuncture in the treatment of chronic pain. Best Pract Res Clin Anaesthesiol. 2020 Sep;34(3):603-616. doi: 10.1016/j.bpa.2020.08.005. Epub 2020 Aug 8. PMID 33004170
- [Background] Lua, P. L., & Talib, N. S. (2012). The effectiveness of auricular acupuncture for drug addiction: a review of research evidence from clinical trials. ASEAN Journal of Psychiatry, 13(1), 55-68.
- [Background] Romoli, M. Ear acupuncture: historical abstract-differences of ear cartography between the east and the west. Dtsch. Z. Akupunkt. 53: 24-33, 2010.
- [Background] Stuyt EB, Voyles CA. The National Acupuncture Detoxification Association protocol, auricular acupuncture to support patients with substance abuse and behavioral health disorders: current perspectives. Subst Abuse Rehabil. 2016 Dec 7;7:169-180. doi: 10.2147/SAR.S99161. eCollection 2016. PMID 27994492
- [Background] Niemtzow, R.C., Battle- field acupuncture. Med. Acupunct. 19: 225-228, 2007.
- [Background] Montgomery AD, Ottenbacher R. Battlefield Acupuncture for Chronic Pain Management in Patients on Long-Term Opioid Therapy. Med Acupunct. 2020 Feb 1;32(1):38-44. doi: 10.1089/acu.2019.1382. Epub 2020 Feb 3. PMID 32110262
- [Background] Lin LL, Li HP, Yang JW, Hao XW, Yan SY, Wang LQ, Yu FT, Shi GX, Liu CZ. Acupuncture for Psychological Disorders Caused by Chronic Pain: A Review and Future Directions. Front Neurosci. 2021 Jan 27;14:626497. doi: 10.3389/fnins.2020.626497. eCollection 2020. PMID 33584181
- [Background] Huang KW, Ochandarena NE, Philson AC, Hyun M, Birnbaum JE, Cicconet M, Sabatini BL. Molecular and anatomical organization of the dorsal raphe nucleus. Elife. 2019 Aug 14;8:e46464. doi: 10.7554/eLife.46464. PMID 31411560
- [Background] Smith MO, Khan I. An acupuncture programme for the treatment of drug-addicted persons. Bull Narc. 1988;40(1):35-41. PMID 3219455
- [Background] Mao JJ, Liou KT, Baser RE, Bao T, Panageas KS, Romero SAD, Li QS, Gallagher RM, Kantoff PW. Effectiveness of Electroacupuncture or Auricular Acupuncture vs Usual Care for Chronic Musculoskeletal Pain Among Cancer Survivors: The PEACE Randomized Clinical Trial. JAMA Oncol. 2021 May 1;7(5):720-727. doi: 10.1001/jamaoncol.2021.0310. PMID 33734288
- [Background] Levy CE, Casler N, FitzGerald DB. Battlefield Acupuncture: An Emerging Method for Easing Pain. Am J Phys Med Rehabil. 2018 Mar;97(3):e18-e19. doi: 10.1097/PHM.0000000000000766. No abstract available. PMID 28570280
- [Background] Vickers AJ, Cronin AM, Maschino AC, Lewith G, MacPherson H, Foster NE, Sherman KJ, Witt CM, Linde K; Acupuncture Trialists' Collaboration. Acupuncture for chronic pain: individual patient data meta-analysis. Arch Intern Med. 2012 Oct 22;172(19):1444-53. doi: 10.1001/archinternmed.2012.3654. PMID 22965186
- [Background] Richard C. Niemtzow.Battlefield Acupuncture.Medical Acupuncture.Dec 2007.225- 228.http://doi.org/10.1089/acu.2007.0603
- [Background] Litscher G. Ear Acupuncture according to the NADA (National Acupuncture Detoxification Association). Medicines (Basel). 2019 Mar 31;6(2):44. doi: 10.3390/medicines6020044. PMID 30935106
- [Background] Garland EL, Hudak J, Hanley AW, Nakamura Y. Mindfulness-oriented recovery enhancement reduces opioid dose in primary care by strengthening autonomic regulation during meditation. Am Psychol. 2020 Sep;75(6):840-852. doi: 10.1037/amp0000638. PMID 32915027
- [Background] Carr DJ. The safety of obstetric acupuncture: forbidden points revisited. Acupunct Med. 2015 Oct;33(5):413-9. doi: 10.1136/acupmed-2015-010936. Epub 2015 Sep 11. PMID 26362792
- [Background] Cook KF, Jensen SE, Schalet BD, Beaumont JL, Amtmann D, Czajkowski S, Dewalt DA, Fries JF, Pilkonis PA, Reeve BB, Stone AA, Weinfurt KP, Cella D. PROMIS measures of pain, fatigue, negative affect, physical function, and social function demonstrated clinical validity across a range of chronic conditions. J Clin Epidemiol. 2016 May;73:89-102. doi: 10.1016/j.jclinepi.2015.08.038. Epub 2016 Mar 4. PMID 26952842
- [Background] Boyett B, Wiest K, McLeod LD, Nelson LM, Bickel WK, Learned SM, Heidbreder C, Fudala PJ, Le Moigne A, Zhao Y. Assessment of craving in opioid use disorder: Psychometric evaluation and predictive validity of the opioid craving VAS. Drug Alcohol Depend. 2021 Dec 1;229(Pt B):109057. doi: 10.1016/j.drugalcdep.2021.109057. Epub 2021 Sep 24. PMID 34794061
- [Background] Lee EH. Review of the psychometric evidence of the perceived stress scale. Asian Nurs Res (Korean Soc Nurs Sci). 2012 Dec;6(4):121-7. doi: 10.1016/j.anr.2012.08.004. Epub 2012 Sep 18. PMID 25031113
- [Background] Buysse DJ, Yu L, Moul DE, Germain A, Stover A, Dodds NE, Johnston KL, Shablesky-Cade MA, Pilkonis PA. Development and validation of patient-reported outcome measures for sleep disturbance and sleep-related impairments. Sleep. 2010 Jun;33(6):781-92. doi: 10.1093/sleep/33.6.781. PMID 20550019
- [Background] Mayer JD, Gaschke YN. The experience and meta-experience of mood. J Pers Soc Psychol. 1988 Jul;55(1):102-11. doi: 10.1037//0022-3514.55.1.102. PMID 3418484
- [Background] Tanay G, Bernstein A. State Mindfulness Scale (SMS): development and initial validation. Psychol Assess. 2013 Dec;25(4):1286-99. doi: 10.1037/a0034044. Epub 2013 Sep 23. PMID 24059475
- [Background] Unintentional Drug Poisoning (Overdose) Deaths in New York City in 2022. Data Brief and Tables, September 2023, No. 137. NYC Office of Chief Medical Examiner and NYC DOHMH Bureau of Vital Statistics, 2000-2022.

DOCUMENTS (1):
  • Informed Consent Form (2025-04-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT06543355/ICF_000.pdf